CLINICAL TRIAL: NCT01090401
Title: PME/Master Study of the Linoxsmart S DX ICD Leads
Brief Title: Linox Smart S DX PME/Master Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Biotronik SE & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 48-1
Record Dates: First submitted 2010-03-18; First posted 2010-03-22 (Estimated); Last update posted 2011-11-16 (Estimated); Status verified 2011-11

CONDITIONS: ICD Indication

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Patients with Linox smart S DX lead (Experimental)
  Interventions: Device: Linox smart S DX

INTERVENTIONS:
Device: Linox smart S DX — ICD lead

SUMMARY:
The objective of this study is to prove the safety and efficacy of the Linox smart S DX ICD lead.

ELIGIBILITY:
Inclusion Criteria:

* Patients with standard ICD indication
* Be available for follow-up visits on a regular basis at an approved investigational center

Exclusion Criteria:

* Patients with standard ICD contra-indication
* Patients with permanent atrial fibrillation
* Have a life expectancy of less than six months
* Are expecting to receive cardiac surgery within 6 months after enrollment
* Age < 18 years
* Not enrolled in another cardiac clinical investigation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2010-03; Primary Completion 2010-12 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Rate of atrial adequate sensing | 6 months

SECONDARY OUTCOMES:
Linox smart S DX related complication-free rate | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Charité University Hospital Benjamin Franklin, Berlin, Germany